CLINICAL TRIAL: NCT06949748
Title: UNIFLECA Study: Prospective Cohort Study on Flecainide's Impact on Persistent High Premature Ventricular Contraction Burden and PVC-Induced Cardiomyopathy
Brief Title: Flecainide in Idiopathic Premature Ventricular Contractions and Related Cardiomyopathy
Acronym: UNIFLECA
Status: Recruiting | Type: Observational
Sponsor: University of Athens (Other)
Collaborators: Institute for Study, Research, Education and Therapy of Vascular, Heart, Brain and Kidney Nosologies (Unknown); University of Patras (Other); University of Crete Medical School - University Hospital of Heraklion (Unknown); Aristotle University Of Thessaloniki (Other); Uni-Pharma (Industry)
Responsible Party: Principal Investigator, Tsiachris Dimitrios, MD, PhD, Assistant Professor of Cardiology, University of Athens
Other Study IDs: 8014/25-04-2024
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Premature Ventricular Beats; Premature Ventricular Complexes; Premature Ventricular Contraction (PVC); Arrhythmia Ventricular; Ventricular Dysfunction, Left; Ventricular Dysfunction; Cardiomyopathies, Secondary; Cardiomyopathies
Keywords: Flecainide; Sanocard; UNIFLECA; PVC induced CMP; PVC; Premature Ventricular Contraction; Outflow Tract PVC; NonOutflow Tract PVC
MeSH Terms: conditions — Ventricular Premature Complexes; Ventricular Dysfunction, Left; Ventricular Dysfunction; Cardiomyopathies | interventions — Flecainide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- High PVC Burden Cohort: Persistent, high PVC Burden (>5%) in 24h Holter Monitoring
  Interventions: Drug: Flecainide (monotherapy)

INTERVENTIONS:
Drug: Flecainide (monotherapy) — • Medication: Flecainide acetate, administered orally.
  * Initial Dosing and Titration:
  * Patients were started on an appropriate dose based on body weight and renal function.
  * The typical starting dose was 100-150 mg per day, split into two doses.
  * Dosing was titrated as needed, depending on patient response and tolerability, under close ECG and clinical monitoring.
  * Monitoring Protocol:
  * Continuous ECG monitoring during drug initiation (especially in-hospital or via Holter).
  * Regular outpatient follow-up visits, including:
  * 12-lead ECGs
  * Holter monitoring
  * Echocardiography (to monitor LVEF and assess for reverse remodeling)
  * ECG parameters (QRS width, QTc interval) were closely monitored for proarrhythmic changes.

SUMMARY:
The UNIFLECA study is a prospective, single-arm, observational cohort evaluating the efficacy, safety, and tolerability of flecainide (in the form of Sanocard) in adults with frequent idiopathic premature ventricular contractions (PVCs) and suspected PVC-induced cardiomyopathy (PVCi-CMP). Frequent PVCs-defined as a burden >5% on two separate 24-hour Holter recordings-are increasingly recognized as a cause of reversible systolic dysfunction in patients without structural heart disease.

Participants undergo a comprehensive baseline evaluation including echocardiography, occasionally cardiac MRI, and coronary angiography or equivalent testing to confirm the absence of structural abnormalities. Patients are enrolled only if they are ineligible or unwilling to undergo catheter ablation, and have no contraindications to flecainide.

Flecainide therapy is initiated at a starting dose of 100 mg/day and titrated up to 200 mg/day, guided by ECG findings, symptom response, and QRS duration. Regular follow-up occurs at three-month intervals over three years, with periodic 24-hour Holter monitoring and assessment of symptoms, LVEF, and adverse events.

The primary outcome is the reduction in PVC burden. Secondary outcomes include improvement in LVEF, symptom relief (measured by structured questionnaires), adverse effects, and long-term treatment adherence. The study aims to generate real-world data on the non-invasive management of PVCs with flecainide and explore its role as an alternative to ablation in carefully selected patients.

DETAILED DESCRIPTION:
The UNIFLECA study is a prospective, single-arm, non-randomized observational cohort designed to evaluate the long-term efficacy and safety of flecainide (in the form of Sanocard) in adult patients with frequent idiopathic premature ventricular contractions (PVCs) and suspected PVC-induced cardiomyopathy (PVCi-CMP). Despite being considered benign in structurally normal hearts, a persistently high PVC burden-particularly above 10%-is increasingly recognized as a cause of reversible left ventricular dysfunction and a potential trigger for cardiomyopathy. This condition is frequently underdiagnosed and may lead to unnecessary treatments or delayed intervention.

The study targets a unique population: symptomatic patients with idiopathic PVCs who have structurally normal hearts and have either declined catheter ablation or are ineligible for invasive procedures. Each patient undergoes comprehensive baseline cardiac evaluation, including transthoracic echocardiography, cardiac magnetic resonance imaging (CMR) to exclude late gadolinium enhancement or myocardial scar, and coronary angiography or non-invasive equivalent to rule out ischemic heart disease. Two 24-hour Holter ECG recordings, taken at least 30 days apart, are used to confirm persistent high PVC burden (>5%).

Flecainide, a Class IC antiarrhythmic agent with sodium channel-blocking properties, is administered as monotherapy. The initial dose is 100 mg/day and may be titrated up to 200 mg/day based on clinical response, patient tolerability, and QRS interval monitoring. Beta-blockers are discontinued unless used for unrelated comorbidities such as hypertension. Patients are monitored with serial 12-lead ECGs, Holter recordings, and echocardiograms at baseline and every three months over a total follow-up period of three years.

The primary endpoint is the percentage reduction in PVC burden as measured by 24-hour Holter ECG. Secondary endpoints include (1) improvement in left ventricular ejection fraction (LVEF), (2) symptom relief as assessed by structured patient questionnaires focusing on palpitations, bradysphygmia, fatigue, dizziness, and exercise intolerance, (3) incidence of adverse events including proarrhythmia, conduction disturbances, and neurological side effects, and (4) adherence to long-term flecainide therapy, including need for dose modifications or drug discontinuation.

This investigator-initiated study is being conducted across tertiary arrhythmia centers in Greece. It aims to fill a significant evidence gap in the long-term pharmacologic management of idiopathic PVCs and PVCi-CMP. Preliminary results indicate significant PVC burden reduction and symptomatic improvement, supporting the potential utility of flecainide as an effective non-invasive therapeutic option in appropriately selected patients. Data from this study will contribute to optimizing treatment strategies for idiopathic ventricular arrhythmias in the absence of structural heart disease, supporting the use of personalized medicine and risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* Frequent idiopathic PVCs (burden >5% on multiple 24-hour Holter ECG recordings)
* Normal cardiac structure and function on echocardiography
* No late gadolinium enhancement or myocardial scar on cardiac MRI
* Normal coronary angiography (excluding ischemic cardiomyopathy)
* Normal serum electrolytes and renal function
* Willingness to comply with follow-up schedule and drug titration

Exclusion Criteria:

* Structural heart disease
* Ischemic heart disease (confirmed by angiography)
* History of sustained ventricular arrhythmias
* Left ventricular ejection fraction (LVEF) <40% at baseline
* Brugada syndrome, long QT syndrome, or other channelopathies
* Contraindications to class IC agents
* Use of concurrent antiarrhythmics or proarrhythmic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population in the UNIFLECA trial consisted of adult patients with frequent idiopathic premature ventricular contractions (PVCs), defined by a PVC burden greater than 5% on multiple 24-hour Holter monitoring. All participants had structurally normal hearts, confirmed by comprehensive imaging including echocardiography, cardiac MRI if necessary, and coronary angiography to exclude cardiomyopathy or ischemic heart disease.
  Eligible individuals were required to have no contraindications to flecainide therapy and no history of sustained ventricular arrhythmias, significant conduction abnormalities, or inherited channelopathies. Patients were selected based on the presence of symptoms such as palpitations or fatigue and a clinical suspicion of PVC-induced cardiomyopathy, without the use of other antiarrhythmic drugs.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
PVC Burden Reduction | 3 years
  Change in 24-hour Holter-measured PVC burden from baseline to 3 years. Unit of Measure: Percent (%)

SECONDARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | 3 years
  * Measured by echocardiography.
  * Unit: Percent (%)
Safety and tolerability of flecainide | 3 years
  * Incidence of adverse effects (e.g., proarrhythmia, dizziness).
  * Unit: Number of participants with event
Symptom improvement (Questionnaire Score) | 3 years
  • Structured patient-reported symptom score (palpitations, fatigue, etc.). • Unit: Score on scale (e.g., 0-10)
Treatment Adherence and Dose Adjustments | 3 years
  * Rate of dose changes or discontinuation due to side effects.
  * Unit: Number of participants

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Tsiachris, MD, PhD, Study Chair — University of Athens
Locations (6):
- Greece (6):
  - Cardiology Clinic, University Hospital of Patras, Pátrai, Achaia
  - 1st Cardiology Clinic, National and Kapodistrian University of Athens, Athens, Attica
  - Cardilogy Clinic, University of Crete, Heraklion
  - 2nd Cardiology Clinic, University of Ioannina, Ioannina
  - 2nd Cardiology Clinic, Aristotle University of Thessaloniki, Thessaloniki
  - 3rd Cardiology Clinic, Aristotle University of Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: No